CLINICAL TRIAL: NCT07280936
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-2906 Injection in Healthy Subjects With a Single Dose and in Obese Patients With Multiple Doses
Brief Title: A Phase I Study of SHR-2906 Injection in Healthy Subjects With a Single Dose and in Obese Patients With Multiple Doses
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2906-101
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2906 Injection Group (Experimental)
  Interventions: Drug: SHR-2906 Injection
- SHR-2906 Injection Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-2906 Injection Placebo

INTERVENTIONS:
Drug: SHR-2906 Injection — SHR-2906 injection, in different doses.
  Arms: SHR-2906 Injection Group
Drug: SHR-2906 Injection Placebo — SHR-2906 injection placebo.
  Arms: SHR-2906 Injection Placebo Group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, dose-escalation phase I clinical trial. This study consists of two parts: the single-dose escalation study (SAD) in healthy subjects and the multiple-dose escalation study (MAD) in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to any study-related activities, understand the procedures and methods of the study, and agree to complete this study in strict accordance with the clinical study protocol;
2. Males or females aged 18-55 years (inclusive);
3. Subjects who are generally healthy as judged by the investigator based on medical history, vital signs, physical examination, laboratory tests, and electrocardiogram (ECG);
4. At screening, 19.0 ≤ BMI ≤ 23.9 kg/m2 (inclusive) for Part I or 28.0 ≤ BMI ≤ 35.0 kg/m2 (inclusive) for Part II.

Exclusion Criteria:

1. During screening, electrocardiogram (ECG) indicated that QTcF>450 ms in males and QTcF> 470 ms in females, as well as other abnormal ECG and vital signs that were judged by the researchers to have clinical significance;
2. There are endocrine diseases or medical histories that may significantly affect body weight during screening (such as Cushing's syndrome, diabetes, hypothyroidism or hyperthyroidism, etc.);
3. There is a history or family history of medullary thyroid carcinoma, multiple endocrine adenomatosis type 2, or a history of pancreatitis or symptomatic gallbladder disease;
4. Other clinical findings within 12 months prior to screening that show clinical significance in the following diseases (including but not limited to gastrointestinal, kidney, liver, nervous, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases);
5. Use of prescription drugs (excluding topical eye/nasal drops and creams without systemic exposure risk), over-the-counter drugs, food supplements, vitamins and Chinese herbal medicines (excluding conventional vitamins) within two weeks prior to screening;
6. Having undergone gastrointestinal surgery that may cause malabsorption before screening, or having taken drugs that directly affect gastrointestinal peristalsis for a long time. For example: having undergone bariatric surgery or procedures (such as gastric banding), or having used weight-reducing drugs (including but not limited to orlistat) within 3 months before administration, or having a weight change of more than 10% within 3 months before administration;
7. Those who have a history of drug abuse in the past five years or have used drugs in the three months prior to the trial; Or the urine drug screening is positive;
8. Blood donation of ≥200 mL within one month prior to screening; Or those who have donated ≥400 mL of blood or lost ≥400 mL of blood within 3 months prior to screening due to trauma or major surgical operations;
9. Inability to tolerate venipuncture for blood collection or fainting at the sight of needles and blood;
10. There are special dietary requirements and they cannot follow the uniform diet;
11. Subjects who the researchers consider to have other factors that make them unsuitable for participating in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs). | Part1: 57 days; Part2: 113 days.
Incidence of serious adverse events (SAEs). | Part1: 57 days; Part2: 113 days.

SECONDARY OUTCOMES:
Maximum concentration (Cmax). | Part1: 57 days; Part2: 113 days.
Time of maximum concentration (Tmax). | Part1: 57 days; Part2: 113 days.
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last). | Part1: 57 days; Part2: 113 days.
Area under the concentration-time curve from time zero to infinity (AUC0-inf). | Part1: 57 days; Part2: 113 days.
Area under the concentration-time curve from time zero to the end of the dosing interval tau (AUC0-tau). | Part1: 57 days; Part2: 113 days.
Elimination half-life (t1/2). | Part1: 57 days; Part2: 113 days.
Apparent clearance (CL/F). | Part1: 57 days; Part2: 113 days.
Apparent volume of distribution (Vz/F). | Part1: 57 days; Part2: 113 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided